CLINICAL TRIAL: NCT00871117
Title: Immunogenicity and Safety Study of Kinrix® Co-administered With Varivax®
Brief Title: Immunogenicity and Safety of Kinrix + (Measles Mumps Rubella) MMR Vaccine With and Without Varicella Vaccine in Healthy Children 4-6 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 111852
Record Dates: First submitted 2009-03-26; First posted 2009-03-30 (Estimated); Results first posted 2011-02-10 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-06

CONDITIONS: Tetanus; Acellular Pertussis; Diphtheria
Keywords: Co-administration; Immunization; Preschool; Booster
MeSH Terms: conditions — Tetanus; Diphtheria

ARMS (2):
- Kinrix + M-M-R II + Varivax (Experimental): Subjects received at Day 0 one dose of Kinrix, intramuscularly in the deltoid region of the left upper arm, co-administered with one dose of M-M-R II and Varivax each, subcutaneously in the deltoid of the right upper and lower arm, respectively.
  Interventions: Biological: GSK Biologicals'Kinrix®; Biological: Merck and Company's MMRII; Biological: Merck and Company's Varivax
- Kinrix + M-M-R II -> Varivax (Active Comparator): Subjects received at Day 0 one dose of Kinrix, intramuscularly in the deltoid region of the left upper arm, co-administered with one dose of M-M-R II, subcutaneously in the deltoid of the right upper arm. At Day 30 they received one dose of Varivax subcutaneously in the deltoid region of the right upper arm.
  Interventions: Biological: GSK Biologicals'Kinrix®; Biological: Merck and Company's MMRII; Biological: Merck and Company's Varivax

INTERVENTIONS:
Biological: GSK Biologicals'Kinrix® — One dose as intramuscular injection at visit 1
Biological: Merck and Company's MMRII — One dose as subcutaneous injection at visit 1
Biological: Merck and Company's Varivax — One dose as subcutaneous injection at visit 1 or at visit 2

SUMMARY:
The purpose of the study is to evaluate the immunogenicity and safety of Kinrix when co-administered with varicella (Varivax® [varicella virus vaccine live], Merck and Company) and (measles mumps rubella) MMR vaccines, compared to Kinrix co-administered with MMR vaccine alone. Both Kinrix and the second dose of Varivax are indicated in children 4-6 years of age, and there is great potential for the vaccines to be given concurrently. The aim of this trial is to demonstrate that co-administered Varivax does not negatively affect the immunogenicity or reactogenicity of Kinrix.

DETAILED DESCRIPTION:
Subjects 4-6 years of age will be randomized into two groups to receive either Kinrix, Varivax and M-M-RII on day 0 (Group 1) or Kinrix and M-M-RII on day 0 and Varivax at month 1(Group 2).

All subjects in both groups to provide blood samples prior to vaccination on day 0 and at month 1 (for Group 2, blood sampling is prior to vaccination with Varivax).

Duration of the study will be approximately 6 months for each subject with a safety telephone contact 6 months after vaccinations.

ELIGIBILITY:
Inclusion Criteria:

* Subjects for whom the investigator believes that their parents/ guardians can and will comply with the requirements of the protocol.
* A male or female child between 4 and 6 years of age, inclusive.
* Written informed consent obtained from the parent or guardian of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Having received 4 doses of (Diphtheria, Tetanus Acellular Pertussis) DTaP vaccine using Pediarix and/or Infanrix, and 3 doses of poliovirus vaccine using Pediarix and/or (inactivated poliovirus vaccine, Aventis Pasteur) IPOL in the first 2 years of life.
* Previously received 1 dose of M-M-RII and Varivax (separate or combined) in the second year of life.

Exclusion Criteria:

* Use of any investigational or non-registered drug or vaccine other than the study vaccines within 30 days preceding the administration of study vaccines, or planned use during the study period.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or non-investigational product or device.
* History of previous or intercurrent diphtheria, tetanus, pertussis, polio, measles, mumps, rubella or varicella disease, or of vaccination against these diseases given after the second year of life.
* Known exposure to diphtheria, tetanus, pertussis, or polio, prior to vaccination.
* Poliovirus vaccination with one or more doses of (oral polio virus) OPV vaccine.
* Administration or planned administration of a vaccine not foreseen by the study protocol within 30 days of study vaccination and ending at Day 30.
* Chronic administration or planned administration of immunosuppressants or other immune modifying drugs within six months prior to study vaccination or planned administration during the study period ending at Day 30.
* Administration of immunoglobulins and/or any blood products at any time prior to study vaccination or planned administration during the study period ending at Day 30.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
* History of seizures or progressive neurological disorder, including infantile spasms, uncontrolled epilepsy or progressive encephalopathy.
* Major congenital defects or serious chronic illness.
* Acute disease at the time of enrolment.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine(s).
* History of anaphylactic reaction to egg proteins or previous doses of the vaccine(s).
* Encephalopathy within 7 days of administration of previous dose of Infanrix or Pediarix.
* Fever >=40.5°C or 104.9°F (rectal temperature) (39.5°C or 103.1°F, oral/axillary) within 48 hours of previous dose of Infanrix or Pediarix not due to another identifiable cause.
* Collapse or shock-like state within 48 hours of previous dose of DTaP or DTaP-containing vaccine.
* Persistent, severe, inconsolable screaming or crying lasting ³3 hours occurring within 48 hours of administration of previous dose of DTaP or DTaP-containing vaccine.
* Thrombocytopenia following a previous dose of M-M-RII or its component vaccines
* Inability to contact a parent/guardian of the subject by telephone.
* Blood dyscrasias, leukemia, lymphomas or other malignant neoplasms affecting the bone marrow or lymphatic systems.
* Family history of congenital or hereditary immunodeficiency, unless the immune competence of the subject has been demonstrated.
* Residence in the same household as the following persons:
* New-born infants (0-4 weeks of age).
* Pregnant mother/women without documented positive history of chickenpox disease or laboratory evidence of prior varicella vaccination.
* Pregnant women at or beyond 28 weeks gestation regardless of varicella vaccination status or varicella disease history.
* Persons with known immunodeficiency.
* Active untreated tuberculosis.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 478 (Actual)
Dates: Start 2009-03-31; Primary Completion 2010-01-15 (Actual); Study Completion 2010-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (10):
- United States (10):
  - GSK Investigational Site, Antioch, California
  - GSK Investigational Site, Daly City, California
  - GSK Investigational Site, Hayward, California
  - GSK Investigational Site, Redwood City, California
  - GSK Investigational Site, Roseville, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Jose, California
  - GSK Investigational Site, Santa Rosa, California
  - GSK Investigational Site, Vallejo, California
  - GSK Investigational Site, Walnut Creek, California

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Klein NP, Weston WM, Kuriyakose S, Kolhe D, Howe B, Friedland LR, Van Der Meeren O. An open-label, randomized, multi-center study of the immunogenicity and safety of DTaP-IPV (Kinrix) co-administered with MMR vaccine with or without varicella vaccine in healthy pre-school age children. Vaccine. 2012 Jan 11;30(3):668-74. doi: 10.1016/j.vaccine.2011.10.065. Epub 2011 Nov 4. PMID 22064267
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 111852 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111852 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111852 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111852 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111852 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111852 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111852 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 478 subjects were enrolled, but 2 subjects who received a subject number were not vaccinated. Therefore the total amount of subjects used for the analysis was 476.
Period: Overall Study
Arm/Group | Kinrix + M-M-R II + Varivax | Kinrix + M-M-R II -> Varivax
Started | 239 | 237
Completed | 234 | 227
Not Completed | 5 | 10
Not completed — Lost to Follow-up | 5 | 6
Not completed — Other | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Kinrix + M-M-R II + Varivax | Kinrix + M-M-R II -> Varivax | Total
Number analyzed (Participants) | 239 | 237 | 476
Age, Continuous [Mean (Standard Deviation); unit: Years] | 4.2 (0.41) | 4.2 (0.37) | 4.2 (0.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129 | 123 | 252
  Male | 110 | 114 | 224
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African Heritage / African American | 27 | 23 | 50
  American Indian or Alaskan Native | 35 | 33 | 68
  Asian - Central/South Asian Heritage | 7 | 11 | 18
  Asian - East Asian Heritage | 3 | 5 | 8
  Asian - South East Asian Heritage | 13 | 17 | 30
  Native Hawaiian or Other Pacific Islander | 2 | 3 | 5
  White - Arabic / North African Heritage | 1 | 6 | 7
  White - Caucasian / European Heritage | 109 | 107 | 216
  Unspecified | 42 | 32 | 74

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Booster Responses to Diphteria and Tetanus
Description: Anti-diphteria (anti-D) and anti-tetanus (anti-T) booster response was defined as:
  * initially seronegative subjects (sero-) (pre-booster antibody concentration below cut-off of < 0.1 international units per milliliter (IU/mL)) with an increase of at least four times the cut-off one month after vaccination (post-booster antibody concentration ≥0.4 IU/mL)
  * initially seropositive subjects (sero+) (pre-booster antibody concentration ≥0.1 IU/mL) with an increase of at least four times the pre-booster antibody concentration one month after vaccination
Time Frame: One month after Kinrix vaccination (Month 1), prior to Varivax vaccination for Kinrix + M-M-R II -> Varivax Group.
Population: Analysis was performed on the according-to-protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom immunogenicity data were available for antibodies against at least one study vaccine antigen component after vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Kinrix + M-M-R II + Varivax | Kinrix + M-M-R II -> Varivax
Number analyzed (Participants) | 211 | 209
Participants
  Anti-D | 209 | 207
  Anti-T: number analyzed (Participants) | 211 | 208
  Anti-T | 208 | 203
Statistical Analysis 1: Comparison: Kinrix + M-M-R II + Varivax vs Kinrix + M-M-R II -> Varivax; To demonstrate the non-inferiority of DTaP-IPV vaccine co-administered with Varicella and MMR vaccines compared to DTaP-IPV vaccine co-administered with MMR only in terms of diphtheria (D) booster response one month after vaccination with DTaP-IPV vaccine; Test type: Non-Inferiority — Lower limit of the standardized asymptotic 95% confidence interval (CI) for the between-group differences in booster response to diphtheria was greater than or equal to (≥)-10%; Difference in booster response rates = 0.01, 95% CI 2-sided [-2.54 to 2.58]
Statistical Analysis 2: Comparison: Kinrix + M-M-R II + Varivax vs Kinrix + M-M-R II -> Varivax; To demonstrate the non-inferiority of DTaP-IPV vaccine co-administered with Varicella and MMR vaccines compared to DTaP-IPV vaccine co-administered with MMR only in terms of tetanus (T) booster response one month after vaccination with DTaP-IPV vaccine; Test type: Non-Inferiority — Lower limit of the standardized asymptotic 95% CI for the between-group differences in booster response to tetanus was ≥ -10%; Difference in booster response rates = 0.98, 95% CI 2-sided [-1.99 to 4.26]

2. Primary Outcome: Number of Subjects With Anti-pertussis Toxoid (Anti-PT), Anti-filamentous Hemagglutinin (FHA) and Anti-pertactin (Anti-PRN) Booster Responses, Measured in Enzyme-Linked Immunosorbent Assay Units Per Milliliter (EL.U/mL)
Description: anti-PT, anti-FHA and anti-PRN booster response :
  * initially sero- (pre-booster antibody concentration below cut-off < 5.0 EL.U/mL) with increase of at least four times cut-off one month after vaccination (concentration post-booster ≥20.0 EL.U/mL)
  * initially sero+ with pre-booster antibody concentration ≥5.0 EL.U/mL and < 20.0 EL.U/mL with increase of at least four times pre-booster concentration one month post-booster
  * initially sero+ with pre-booster antibody concentration ≥20.0 EL.U/mL with an increase of at least two times the pre-booster antibody concentration one month post-booster
Time Frame: One month after Kinrix vaccination (Month 1), prior to Varivax vaccination for Kinrix + M-M-R II -> Varivax Group.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Kinrix + M-M-R II + Varivax | Kinrix + M-M-R II -> Varivax
Number analyzed (Participants) | 220 | 212
Participants
  Anti-PT: number analyzed (Participants) | 218 | 210
  Anti-PT | 207 | 201
  Anti-FHA: number analyzed (Participants) | 216 | 210
  Anti-FHA | 213 | 209
  Anti-PRN | 220 | 209
Statistical Analysis 1: Comparison: Kinrix + M-M-R II + Varivax vs Kinrix + M-M-R II -> Varivax; To demonstrate the non-inferiority of DTaP-IPV vaccine co-administered with Varicella and MMR vaccines compared to DTaP-IPV vaccine co-administered with MMR only in terms of pertussis toxoid (PT) booster response one month after vaccination with DTaP-IPV vaccine; Test type: Non-Inferiority — Lower limit of the standardized asymptotic 95% CI for the between-group differences in booster response to PT was ≥ -10%; Difference in booster response rates = -0.76, 95% CI 2-sided [-5.07 to 3.51]
Statistical Analysis 2: Comparison: Kinrix + M-M-R II + Varivax vs Kinrix + M-M-R II -> Varivax; To demonstrate the non-inferiority of DTaP-IPV vaccine co-administered with Varicella and MMR vaccines compared to DTaP-IPV vaccine co-administered with MMR only in terms of filamentous hemagglutinin (FHA) booster response one month after vaccination with DTaP-IPV vaccine; Test type: Non-Inferiority — Lower limit of the standardized asymptotic 95% CI for the between-group differences in booster response to FHA was ≥ -10%; Difference in booster response rates = -0.91, 95% CI 2-sided [-3.59 to 1.39]
Statistical Analysis 3: Comparison: Kinrix + M-M-R II + Varivax vs Kinrix + M-M-R II -> Varivax; To demonstrate the non-inferiority of DTaP-IPV vaccine co-administered with Varicella and MMR vaccines compared to DTaP-IPV vaccine co-administered with MMR only in terms of pertactin (PRN) booster response one month after vaccination with DTaP-IPV vaccine; Test type: Non-Inferiority — Lower limit of the standardized asymptotic 95% CI for the between-group differences in booster response to PRN, was ≥ -10%; Difference in booster response rates = 1.42, 95% CI 2-sided [-0.32 to 4.08]

3. Primary Outcome: Geometric Mean Titers (GMTs) for Antibodies to Poliovirus Types 1, 2 and 3
Description: Titers are expressed as GMTs.
Time Frame: One month after Kinrix vaccination (Month 1), prior to Varivax vaccination for Kinrix + M-M-R II -> Varivax Group.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Kinrix + M-M-R II + Varivax | Kinrix + M-M-R II -> Varivax
Number analyzed (Participants) | 219 | 212
titer
  Anti-Polio 1: number analyzed (Participants) | 219 | 211
  Anti-Polio 1 | 1638.4 [1441.0 to 1863.0] | 1789.9 [1559.0 to 2054.9]
  Anti-Polio 2: number analyzed (Participants) | 218 | 212
  Anti-Polio 2 | 1572.9 [1387.8 to 1782.7] | 1902.6 [1678.6 to 2156.5]
  Anti-Polio 3 | 2588.4 [2282.7 to 2935.0] | 3189.6 [2798.2 to 3635.7]
Statistical Analysis 1: Comparison: Kinrix + M-M-R II + Varivax vs Kinrix + M-M-R II -> Varivax; To demonstrate the non-inferiority of DTaP-IPV vaccine co-administered with Varicella and MMR vaccines compared to DTaP-IPV vaccine co-administered with MMR only in terms of poliovirus type 1 geometric mean titers (GMTs), one month after vaccination with DTaP-IPV vaccine; Test type: Non-Inferiority — Lower limit of the 95% CI for the GMT ratios for poliovirus type 1 antigens was ≥ 0.67; Adjusted GMT ratio = 0.91, 95% CI 2-sided [0.76 to 1.1]
Statistical Analysis 2: Comparison: Kinrix + M-M-R II + Varivax vs Kinrix + M-M-R II -> Varivax; To demonstrate the non-inferiority of DTaP-IPV vaccine co-administered with Varicella and MMR vaccines compared to DTaP-IPV vaccine co-administered with MMR only in terms of poliovirus type 2 geometric mean titers (GMTs), one month after vaccination with DTaP-IPV vaccine; Test type: Non-Inferiority — Lower limit of the 95% CI for the GMT ratios of poliovirus type 2 antigens was ≥ 0.67; Adjusted GMT ratio = 0.83, 95% CI 2-sided [0.7 to 0.99]
Statistical Analysis 3: Comparison: Kinrix + M-M-R II + Varivax vs Kinrix + M-M-R II -> Varivax; To demonstrate the non-inferiority of DTaP-IPV vaccine co-administered with Varicella and MMR vaccines compared to DTaP-IPV vaccine co-administered with MMR only in terms of poliovirus type 3 geometric mean titers (GMTs), one month after vaccination with DTaP-IPV vaccine; Test type: Non-Inferiority — Lower limit of the 95% CI for the GMT ratios of poliovirus type 3 antigens was ≥ 0.67; Adjusted GMT ratio = 0.84, 95% CI 2-sided [0.71 to 1.01]

4. Secondary Outcome: Number of Subjects With Anti-D and Anti-T Antibody Concentrations Above Cut-off Value
Description: Cut-off value was defined as greater than or equal to 1.0 international units per milliliter (IU/mL).
Time Frame: One month after Kinrix vaccination (Month 1), prior to Varivax vaccination for Kinrix + M-M-R II -> Varivax Group.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Kinrix + M-M-R II + Varivax | Kinrix + M-M-R II -> Varivax
Number analyzed (Participants) | 217 | 212
Participants
  Anti-D | 217 | 212
  Anti-T | 217 | 209

5. Secondary Outcome: Geometric Mean Concentrations (GMCs) for Anti-D and Anti-T Antibodies
Description: Concentrations were expressed as GMCs in IU/mL.
Time Frame: One month after Kinrix vaccination (Month 1), prior to Varivax vaccination for Kinrix + M-M-R II -> Varivax Group.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Kinrix + M-M-R II + Varivax | Kinrix + M-M-R II -> Varivax
Number analyzed (Participants) | 217 | 212
IU/mL
  Anti-D | 14.273 [12.989 to 15.684] | 14.809 [13.397 to 16.371]
  Anti-T | 8.658 [7.888 to 9.504] | 8.138 [7.323 to 9.045]

6. Secondary Outcome: GMCs for Anti-PT, Anti-FHA, Anti-PRN Antibodies
Description: Concentrations are expressed as GMCs in Enzyme-Linked Immunosorbent Assay (ELISA) Units per milliliter (EL.U/mL).
Time Frame: One month after Kinrix vaccination (Month 1), prior to Varivax vaccination for Kinrix + M-M-R II -> Varivax Group.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Kinrix + M-M-R II + Varivax | Kinrix + M-M-R II -> Varivax
Number analyzed (Participants) | 220 | 212
EL.U/mL
  Anti-PT | 96.5 [85.8 to 108.6] | 101.3 [89.2 to 115.1]
  Anti-FHA | 968.9 [886.9 to 1058.4] | 968.2 [876.0 to 1070.1]
  Anti-PRN | 627.1 [543.2 to 724.0] | 620.4 [530.3 to 725.8]

7. Secondary Outcome: Number of Subjects With an Anti-polio 1, 2, 3 Booster Response
Description: Anti-poliovirus 1, anti-poliovirus 2 and anti-poliovirus 3 booster response:
  * initially seronegative subjects (pre-booster antibody titer below cut-off of 8 ED50) with an antibody titer ≥ 32 ED50 one month after vaccination
  * initially seropositive subjects (pre-booster antibody titers ≥ 8 ED50) with an increase at least four times the pre-booster antibody titer one month after vaccination.
  ED50 is defined here as the reverse of the dilution resulting in 50% inhibition. The lowest dilution at which serum samples were tested is 1:8 from which a test was considered positive.
Time Frame: One month after Kinrix vaccination (Month 1), prior to Varivax vaccination for Kinrix + M-M-R II -> Varivax Group.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Kinrix + M-M-R II + Varivax | Kinrix + M-M-R II -> Varivax
Number analyzed (Participants) | 215 | 211
Participants
  Anti-polio 1: number analyzed (Participants) | 215 | 209
  Anti-polio 1 | 211 | 202
  Anti-polio 2: number analyzed (Participants) | 214 | 211
  Anti-polio 2 | 204 | 207
  Anti-polio 3 | 213 | 207

8. Secondary Outcome: Number of Subjects Seroprotected Against Diphteria and Tetanus
Description: Seroprotection status was defined as:
  * anti-D antibody concentration greater than or equal to 0.1 IU/mL
  * anti-T antibody concentration greater than or equal to 0.1 IU/mL
Time Frame: One month after Kinrix vaccination (Month 1), prior to Varivax vaccination for Kinrix + M-M-R II -> Varivax Group.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Kinrix + M-M-R II + Varivax | Kinrix + M-M-R II -> Varivax
Number analyzed (Participants) | 217 | 212
Participants
  Anti-D | 217 | 212
  Anti-T | 217 | 212

9. Secondary Outcome: Number of Subjects Protected Against Poliovirus 1, 2 and 3
Description: Seroprotection was defined:
  * anti-poliovirus type 1, 2 or 3 antibody titer greater than or equal to 8 ED50.
  ED50 is defined here as the reverse of the dilution resulting in 50% inhibition.
Time Frame: One month after Kinrix vaccination (Month 1), prior to Varivax vaccination for Kinrix + M-M-R II -> Varivax Group.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Kinrix + M-M-R II + Varivax | Kinrix + M-M-R II -> Varivax
Number analyzed (Participants) | 219 | 212
Participants
  Anti-Polio 1: number analyzed (Participants) | 219 | 211
  Anti-Polio 1 | 219 | 211
  Anti-Polio 2: number analyzed (Participants) | 218 | 212
  Anti-Polio 2 | 218 | 212
  Anti-Polio 3 | 219 | 212

10. Secondary Outcome: Number of Subjects Seropositive for Anti-PT, Anti-FHA and Anti-PRN Antibodies
Description: Seropositivity was defined as a concentration greater than or equal to 5.0 EL.U/mL
Time Frame: One month after Kinrix vaccination (Month 1), prior to Varivax vaccination for Kinrix + M-M-R II -> Varivax Group.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Kinrix + M-M-R II + Varivax | Kinrix + M-M-R II -> Varivax
Number analyzed (Participants) | 220 | 212
Participants
  anti-PT | 220 | 212
  anti-FHA | 220 | 212
  anti-PRN | 220 | 212

11. Secondary Outcome: Number of Subjects With Any Solicited Local Symptoms
Description: Solicited local symptoms included pain, redness and swelling at the injection site. Any was defined as incidence of a particular symptom regardless of intensity grade.
Time Frame: Within 4 days (Day 0 to 3) after booster immunization * for Kinrix + M-M-R II -> Varivax Group before vaccination with Varivax
Population: The analysis was performed on the total vaccinated cohort, which included subjects with at least one vaccine administration documented, only on subjects with their symptom sheets completed.
Measure: Count of Participants; unit: Participants
Groups:
- Kinrix + M-M-R II -> Varivax: Subjects received at Day 0 one dose of Kinrix,intramuscularly in the deltoid region of the left upper arm, co-administered with one dose of M-M-R II, subcutaneously in the deltoid of the right upper arm. At Day 30 they received one dose of Varivax subcutaneously in the deltoid region of the right upper arm.
Arm/Group | Kinrix + M-M-R II + Varivax | Kinrix + M-M-R II -> Varivax
Number analyzed (Participants) | 230 | 230
Participants
  Any Pain | 156 | 166
  Any Redness | 115 | 114
  Any Swelling | 95 | 84

12. Secondary Outcome: Number of Subjects With Any Solicited General Symptoms
Description: Solicited general symptoms included fever [temperature equal to or greater than 37.5 degrees Celsius (°C)], drowsiness and loss of appetite. Any was defined as incidence of a particular symptom regardless of intensity grade.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Kinrix + M-M-R II + Varivax | Kinrix + M-M-R II -> Varivax
Number analyzed (Participants) | 230 | 230
Participants
  Any Drowsiness | 61 | 66
  Any Loss of appetite | 60 | 57
  Any Temperature (Axillary) | 58 | 68

13. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events
Description: An unsolicited adverse event is any adverse event (i.e. any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product) reported in addition to those solicited during the clinical study. Also any "solicited" symptom with onset outside the specified period of follow-up for solicited symptoms will be reported as an unsolicited adverse event.
Time Frame: Up to 31 days (Day 0 through Day 30) after booster vaccination * for Kinrix + M-M-R II -> Varivax Group before vaccination with Varivax
Population: Analysis was performed on the total vaccinated cohort, which included all subjects with at least one vaccine administration documented and for whom data was available.
Measure: Count of Participants; unit: Participants
Arm/Group | Kinrix + M-M-R II + Varivax | Kinrix + M-M-R II -> Varivax
Number analyzed (Participants) | 239 | 237
Participants | 75 | 72

14. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events are medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: During the entire study period (from Day 0 to 6 months post-vaccination)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Kinrix + M-M-R II + Varivax | Kinrix + M-M-R II -> Varivax
Number analyzed (Participants) | 239 | 237
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: Solicited local/general Adverse Events (AEs) during the first 4 days (Day 0-3) post vaccination ; unsolicited AEs during the 31 days (Days 0-30) post vaccination and SAEs during the entire study period (from Day 0 to 6 months post-vaccination).
Description: Solicited local/general Adverse Events (AEs) were only collected from subjects with their symptom sheets completed.
Groups:
- Kinrix + M-M-R II + Varivax: Subjects received at Day 0 one dose of Kinrix,intramuscularly in the deltoid region of the left upper arm, co-administered with one dose of M-M-R II, subcutaneously in the deltoid of the right upper arm, and one dose of Varivax subcutaneously in the deltoid region of the right lower arm.
Arm/Group | Kinrix + M-M-R II + Varivax | Kinrix + M-M-R II -> Varivax
All-Cause Mortality (participants affected / at risk) | 0/239 | 0/237
Serious Adverse Events (participants affected / at risk) | 0/239 | 1/237
Other Adverse Events (participants affected / at risk) | 228/230 | 230/230
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Kinrix + M-M-R II + Varivax (N=239) | Kinrix + M-M-R II -> Varivax (N=237)
Croup infectious (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Kinrix + M-M-R II + Varivax (N=230) | Kinrix + M-M-R II -> Varivax (N=230)
Pain (General disorders) | 156 | 166 — This solicited local symptom was only collected from subjects with their symptom sheets completed.
Redness (General disorders) | 115 | 114 — This solicited local symptom was only collected from subjects with their symptom sheets completed.
Swelling (General disorders) | 95 | 84 — This solicited local symptom was only collected from subjects with their symptom sheets completed.
Drowsiness (General disorders) | 61 | 66 — This solicited general symptom was only collected from subjects with their symptom sheets completed.
Loss of appetite (General disorders) | 60 | 57 — This solicited general symptom was only collected from subjects with their symptom sheets completed.
Fever (General disorders) | 58 | 68 — This solicited general symptom was only collected from subjects with their symptom sheets completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.